CLINICAL TRIAL: NCT04043793
Title: Intensive Care Unit (ICU)-Acquired Colonization and Infection Related to Multidrug Resistant Bacteria (MDR) in Immunocompromised Patients
Brief Title: ICU-acquired Colonization and Infection Related to MDR in Immunocompromised Patients
Acronym: CIMDREA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_07; 2018-A02756-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-07-03; First posted 2019-08-02 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Immunocompromised Host; Critical Care
Keywords: Immunocompromised Host; Critical care; Drug Resistance, Multiple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the number of immunocompromised patients hospitalized in the intensive care units (ICU) is increasing. They are at higher risk of colonization and/or infection with multi-resistant bacteria (MDR). However this risk is not well characterized. ICU acquired infections related to MDR are associated with increased morbidity and mortality. The aim of this study is to compare the incidence of ICU-acquired colonization and ICU-acquired infection related to MDR between immunocompromized and immunocompetent patients. The risk factors for ICU-acquired colonization and ICU-acquired infections, and their impact on outcome will also be evaluated and compared between immunocompromised and immunocompetent patients.

ELIGIBILITY:
Inclusion Criteria:

* Expected ICU stay > 48 hours
* All patients (immunocompromised or immunocompetent).

Exclusion Criteria:

* Patients aged < 18 years
* Refusal to take part in the study
* ICU-stay < 48 hours
* Non availability of initial MDR or subsequent screening
* Participation in another study that could interfere with the risk of ICU-acquired colonization and infection with MDR bacteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: immunocompetent patients, and immunocompromised patients admitted to intensive care
Sampling Method: Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Density rate of ICU-acquired infections related to MDR in immunosuppressed patients. | From ICU admission until day 28 after ICU admission
  the number ICU-acquired infections related to MDR will be devided by the number of days in the ICU and reported for 1000 days.

SECONDARY OUTCOMES:
Density rate of ICU-acquired colonizations related to MDR in immunosuppressed patients | From ICU admission until day 28 after ICU admission
  the number of ICU-acquired colonizations related to MDR will be devided by the number of days in the ICU and reported for 1000 days
Rate of ICU-acquired colonizations related to MDR in immunosuppressed patients. | From ICU admission until day 28 after ICU admission
  The rate of patients with at least one ICU-acquired colonization related to MDR
Rate of ICU-acquired infections related to MDR in immunosuppressed patients | From ICU admission until day 28 after ICU admission
  The rate of patients with at least one ICU-acquired infection related to MDR
28 day mortality | from ICU admission until day 28 after admission
  death in the ICU or after discharge from the ICU
Mechanical ventilation duration | From ICU admission until day 28 after ICU admission
  the number of days Under mechanical ventilation
length of stay in intensive care unit | From ICU admission until day 28 after ICU admission
  the number of days of hospitalization in teh ICU

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Chu Amiens Picardie, Amiens
  - Ch Bethune, Béthune
  - Grand Hopital de L'Est Francilien, Jossigny
  - CH LENS, Lens
  - Hôpital Roger Salengro, CHU, Lille
  - Hospices Civils de Lyon, Lyon
  - C.H de Roubaix, Roubaix